CLINICAL TRIAL: NCT02661373
Title: Phase 1a, First-In-Human, Dose-Escalation Study of (+)-SJ000557733 (SJ733), an Oral, Novel Inhibitor of Plasmodium Falciparum Plasma Membrane Protein PfATP4
Brief Title: First-in-Human Study of an Oral Plasmodium Falciparum Plasma Membrane Protein Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Medicines for Malaria Venture (Other); Eisai Inc. (Industry); Global Health Innovative Technology Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BUZZOFF
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Malaria
Keywords: Antimalarial; First-in-Human; Pharmacokinetic
MeSH Terms: conditions — Malaria | interventions — SJ733; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants will receive SJ733, an investigational drug developed at St. Jude Children's Research Hospital, and cobicistat.
  Interventions: Drug: SJ733; Drug: Cobicistat

INTERVENTIONS:
Drug: SJ733 — SJ733 is an oral, novel inhibitor of Plasmodium Falciparum plasma membrane protein PFATP4. It will be administered as a single, multi, or boosted oral dose.
  Other Names: (+)-SJ000557733
Drug: Cobicistat — Commercially available cobicistat 150 mg tablets will be used. It will be administered as a single oral dose together with SJ733.
  Other Names: Tybost®

SUMMARY:
Malaria is an infectious disease caused by a parasite that is passed to humans when an infected mosquito bites a person. About 3.4 billion people live in areas of the world where malaria is regularly found. In many countries, malaria is one of the leading causes of illness and death. Despite this, there are a limited number of drugs, called antimalarials, that can be used to treat malaria and increasing reports of resistance to existing antimalarials.

The purpose of this research study is to test a new experimental antimalarial drug called SJ733 to first assess its safety, tolerability and blood levels in healthy adult volunteers.

Single-dose, multi-dose and boosted-dose cohorts (both single and multi-dose) will be studied. The pharmacoenhancer (booster), cobicistat, will be given in combination with SJ733 in the boosted dose-cohorts.

PRIMARY OBJECTIVES:

* To assess the preliminary safety and tolerability of escalating doses of antimalarial SJ733 in healthy human volunteers.
* To investigate the pharmacokinetic (PK) profile of escalating doses of antimalarial SJ733 and its metabolite in healthy human volunteers.
* To identify a dose of SJ733 that can be tested in a separate Phase 1b human malaria challenge study.
* To assess the preliminary safety and tolerability of SJ733 in healthy adult volunteers after multiple oral dosing.
* To assess the pharmacokinetics of SJ733 and its metabolite SJ506 after multiple dosing of SJ733 in healthy adult volunteers.
* To assess the preliminary safety and tolerability of escalating single oral doses of SJ733 in combination with cobicistat among healthy adult volunteers.
* To assess the pharmacokinetics of SJ733 and its metabolite SJ506 after single oral doses of SJ733 in combination with cobicistat among healthy adult volunteers.
* To assess the preliminary safety and tolerability of SJ733 in combination with cobicistat in healthy adult volunteers after multiple oral dosing.
* To assess the pharmacokinetics of SJ733 and its metabolite SJ506 after multiple dosing of SJ733 in combination with cobicistat among healthy volunteers.

SECONDARY OBJECTIVE:

* To assess the impact of food intake on the pharmacokinetic profile of antimalarial SJ733.

DETAILED DESCRIPTION:
This is a single site, Phase 1a, first-in-human, oral, primarily single-dose, dose escalation study of (+)-SJ000557733 (SJ733) in healthy adult volunteers. SJ733, is an investigational oral anti-malarial agent is a novel inhibitor of Plasmodium falciparum plasma membrane protein (PfATP4). Subjects meeting eligibility criteria will be enrolled using a leap frog, fixed dose escalation design with an adaptive component where 6 subjects are enrolled per dose cohort.

Following successful completion of the safety and pharmacokinetic (PK) assessment resulting from the single-dose escalation portion of the study, a three-dose cohort study will be undertaken. It includes once per day oral dosing for 3 consecutive days. Both single and multi-dose cohorts of SJ733 in combination with cobicistat (boosted cohorts) will also be completed.

After the study results from the single-dose cohorts of SJ733 in combination with cobicistat (boosted cohorts) were reviewed, multi-dose cohorts of SJ733 in combination with cobicistat (boosted cohorts) were not conducted and Phase 2 study planning initiated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (as certified by comprehensive medical assessment including detailed history and complete physical examination), male or female, aged 18 to 55 years of age (inclusive) at screening
* At least 50 kg in weight and body mass index (BMI) between 18 and 34 kg/m^2
* Able and willing to provide informed consent and to be available for follow-up for the planned duration of the study
* If female, then not of child bearing potential (i.e. permanently sterilized hysterectomy or bilateral oophorectomy at least 6 months before screening; proper documentation required] and/or post-menopausal defined as 12 months with no menses without an alternative cause and with an estradiol level of < 30 pg/mL and follicle-stimulating hormone level of > 40 IU/L at screening)
* Sexually active males must agree to be abstinent or use condoms for the duration of the study.
* Screening laboratories (hematology, chemistries, venous methemoglobin level specified in schedule of evaluations) within normal institutional range or if outside the range, not clinically significant in the opinion of the investigator.

Inclusion Criteria for Participants in Single-dose Cohort Only::

* Agrees not to receive any vaccination within 7 days prior to Day 0 and through Day 7.
* Agrees not to use nonprescription drugs, including vitamins, antacids, and herbal and dietary supplements within 7 days prior to Day 0 and through Day 7. Acetaminophen may be used at doses of ≤ 1 g/day, and ibuprofen may be used at doses of ≤ 1.2 g/day.
* Agrees not to use nicotine containing products from screening through Day 7.
* Agrees not to consume alcohol for the 24 hours prior to Day 0 and through Day 7.
* Agrees not to eat pomegranate, grapefruit or other citrus fruits or drink their juices within 7 days prior to Day 0 and through Day 7.
* Agrees to limit caffeine to no more than 200 mg on Day 0.
* Agrees not to eat or drink (except water) for 10 hours before the Day 0 visit and have no water for the hour prior to dosing.

Exclusion Criteria:

* Presence of a significant medical or psychiatric condition that in the opinion of the investigator precludes participation in the study.
* Clinically significant abnormalities on physical examination that, in the opinion of the investigator, would preclude entry into the study.
* History of having a significant illness within the 2 weeks prior to screening visit. Participants can screen after illness is resolved for two weeks.
* History of clinically significant electrocardiogram abnormalities or clinically significant abnormalities from the screening electrocardiogram.
* G6PD deficiency
* History of hemolytic anemia or methemoglobinemia
* History of severe drug hypersensitivity including a severe allergic reaction, anaphylaxis or convulsions following any medication, vaccination or infusion.
* History of drug or alcohol abuse in the 12 months prior to screening or evidence at screening visit
* Use of nicotine containing products within 30 days prior to screening
* Positive blood test for HBsAg, HCV, or HIV-1
* Participation in a clinical study of another investigational product within 30 days prior to study enrollment, or planning to begin such participation during the study.
* Employment under the direct supervision of the investigators or study staff.
* Receipt of any vaccination within 7 days of dosing.
* Febrile illness within 48 hours of dosing
* Use of any prescription medication within 14 days prior to study drug administration.
* Use of nonprescription drugs, including vitamins, antacids, and herbal and dietary supplements within 7 days prior to study drug administration. Acetaminophen may be used at doses of ≤ 1 g/day, and ibuprofen may be used at doses of ≤ 1.2 g/day.
* Consumption of pomegranate, grapefruit or other citrus fruits or their juices within 7 days prior to study drug administration.
* Use of nicotine containing products from screening to study drug administration.
* Consumption of alcohol within 24 hours prior to study drug administration.

Inclusion Criteria For participants in multi-dose cohort only:

* Agrees not to receive any vaccination within 7 days prior to Day 1 and through Day 10.
* Agrees not to use nonprescription drugs, including vitamins, antacids, and herbal and dietary supplements within 7 days prior to Day 1 and through Day 10. Acetaminophen may be used at doses of ≤ 1 g/day, and ibuprofen may be used at doses of ≤ 1.2 g/day.
* Agrees not to use nicotine containing products from screening through Day 10.
* Agrees not to consume alcohol for the 24 hours prior to Day 1 and through Day 10.
* Agrees not to eat pomegranate, grapefruit or other citrus fruits or drink their juices within 7 days prior to Day 1 and through Day 10.
* Agrees to limit caffeine to no more than 200 mg on Days 1, 2, and 3.
* Agrees not to eat or drink (except water) for 10 hours before the Days 1, 2, and 3 visits and have no water for the hour prior to dosing on each of those days.

Note: As with the single dose study, sexually active must agree to be abstinent or use condoms for the duration of the study (through the Day 14 visit).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | From baseline up to minimum of 7 days post-dose
  Number of DLT events will be described at each study dose level. DLT is defined as possibly, probably, or definitely related Grade 4 event, possibly, probably or definitely related Grade 3 event, or possibly, probably, or definitely related Grade 2 methemoglobinemia or anemia (attributed to hemolysis) events.
Maximum tolerated dose (MTD) | 7 days after the last dose administration
  MTD is defined as the dose level prior to the dose cohort that 2 or more Grade 2 methemoglobinemia or anemia (attributed to hemolysis) OR any related Grade 3 OR any Grade 4, study drug adverse event (AE) occurred in.
Drug absorption | From baseline through 7 days post-dose
  Drug absorption of SJ733 and its metabolite will be reported.
Drug clearance | From baseline through 7 days post-dose
  Drug clearance of SJ733 and its metabolite will be reported.
Drug volume of distribution | From baseline through 7 days post-dose
  Drug volume of distribution of SJ733 and its metabolite will be reported.
Area under the curve (AUC) | From baseline through 7 days post-dose
  AUC of SJ733 and its metabolite will be reported.
Time above threshold concentration | From baseline through 7 days post-dose
  Time above threshold concentration of SJ733 and its metabolite will be reported.
Maximum drug concentration (Cmax) | From baseline through 7 days post-dose
  Cmax of SJ733 and its metabolite will be reported.
Dose level of SJ733 | 14 days after the last dose administration
  The dose chosen for the phase 1b trial will be no greater than the MTD and provide an exposure (AUC and time above threshold concentration) that equates (using applicable scaling) with those that provided maximum parasitological effect in the gold standard rodent model.

SECONDARY OUTCOMES:
Drug absorption in the fed cohort | From baseline through 7 days post-dose
  Drug absorption of SJ733 and its metabolite in the fed cohort will be reported to assess the impact of food intake.
Drug clearance in the fed cohort | From baseline through 7 days post-dose
  Drug clearance of SJ733 and its metabolite in the fed cohort will be reported to assess the impact of food intake.
Drug volume of distribution in the fed cohort | From baseline through 7 days post-dose
  Drug volume of distribution of SJ733 and its metabolite in the fed cohort will be reported to assess the impact of food intake.
Area under the curve (AUC) in the fed cohort | From baseline through 7 days post-dose
  AUC of SJ733 and its metabolite in the fed cohort will be reported to assess the impact of food intake.
Time above threshold concentration in the fed cohort | From baseline through 7 days post-dose
  Time above threshold concentration SJ733 and its metabolite in the fed cohort will be reported to assess the impact of food intake.
Maximum drug concentration (Cmax) in the fed cohort | From baseline through 7 days post-dose
  Drug absorption of SJ733 and its metabolite in the fed cohort will be reported to assess the impact of food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Aditya H. Gaur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Gaur AH, Panetta JC, Smith AM, Dallas RH, Freeman BB 3rd, Stewart TB, Tang L, John E, Branum KC, Patel ND, Ost S, Heine RN, Richardson JL, Hammill JT, Bebrevska L, Gusovsky F, Maki N, Yanagi T, Flynn PM, McCarthy JS, Chalon S, Guy RK. Combining SJ733, an oral ATP4 inhibitor of Plasmodium falciparum, with the pharmacokinetic enhancer cobicistat: An innovative approach in antimalarial drug development. EBioMedicine. 2022 Jun;80:104065. doi: 10.1016/j.ebiom.2022.104065. Epub 2022 May 19. PMID 35598441
- [Derived] Gaur AH, McCarthy JS, Panetta JC, Dallas RH, Woodford J, Tang L, Smith AM, Stewart TB, Branum KC, Freeman BB 3rd, Patel ND, John E, Chalon S, Ost S, Heine RN, Richardson JL, Christensen R, Flynn PM, Van Gessel Y, Mitasev B, Mohrle JJ, Gusovsky F, Bebrevska L, Guy RK. Safety, tolerability, pharmacokinetics, and antimalarial efficacy of a novel Plasmodium falciparum ATP4 inhibitor SJ733: a first-in-human and induced blood-stage malaria phase 1a/b trial. Lancet Infect Dis. 2020 Aug;20(8):964-975. doi: 10.1016/S1473-3099(19)30611-5. Epub 2020 Apr 8. PMID 32275867
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols